CLINICAL TRIAL: NCT03717454
Title: The Predictive Value of Positron Emission Tomography-Magnetic Resonance (PET-MR) Mediated Dopamine D2 Receptors Imaging in the Drug Therapy of of Prolactinomas.
Brief Title: Dopamine D2 Receptors(D2R) Imaging in Prolactinomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhebao Wu (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); First Hospital of China Medical University (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Peking Union Medical College Hospital (Other); Huashan Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhebao Wu, Principal Investigator, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DD2RP-2018
Record Dates: First submitted 2018-10-14; First posted 2018-10-24 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Prolactinoma
Keywords: Dopamine agonist; Dopamine D2 receptors; PET-MR
MeSH Terms: conditions — Prolactinoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug treatment (Experimental): Subjects are treated with CAB tablets 2mg/week or BC tablets 7.5mg/day.The pituitary hormone levels, tumor volume,visual acuity and visual field scale will be measured every 3 months.MRI showed that the tumors shrunk significantly.
  Interventions: Drug: Drug treatment
- Surgery (Experimental): Subjects are treated with CAB tablets 2mg/week or BC tablets 7.5mg/day.The pituitary hormone levels, tumor volume, visual acuity and visual field scale will be measured every 3 months. The CAB or BC fail to decrease prolactinoma size.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — The medication will be stopped if failure to decrease prolactinoma size and the subjects will be advised to endoscopic transphenoidal pituitary surgery .
  Arms: Surgery
Drug: Drug treatment — The medication will continue if DA causes tumors to shrink.
  Arms: Drug treatment

SUMMARY:
To study the in vivo expression of dopamine D2 receptors in prolactinoma and the predictive role of dopamine D2 receptors PET-MR imaging in the therapeutic effect of dopamine agonists.

DETAILED DESCRIPTION:
The dopamine agonist(DA),such as cabergoline(CAB) and bromocriptine(BC), has been used widely in the treatment of prolactinomas, but its clinical use is hampered by intolerance and/or resistant in some patients. It had been showed that DA inhibit prolactin secretion by binding to and activating dopamine D2 receptors.PET-MR combined MR images with PET function images is substantial to evaluate the expression of dopamine D2 receptors.The aim is to study the in vivo expression of dopamine D2 receptors in prolactinoma and the predictive role of dopamine D2 receptors PET-MR imaging in the therapeutic effect of DA.

ELIGIBILITY:
Inclusion Criteria:

1. Hyperprolactinemia;
2. Enhanced pituitary MRI shows sella regional tumor;
3. Aged between 18 and 65 years old, either sex;
4. Karnofsky performance status ≥ 70;
5. The patient has signed the informed consent.

Exclusion Criteria:

1. Patients concomitantly taking the psychotropic drugs or other drugs causing elevated PRL ;
2. Patients with parkinson disease and is taking dopaminergic agents;
3. Patients with prolactinoma who received Gamma knife treatment;
4. Pregnant or lactating women, or women preparing pregnant;
5. Patients with poor compliance, who cannot implement the program strictly.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabergoline.
7. Patients with claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on PRL level | Up to 6 months
  Record the result of PRL on every 3 month follow-up visit

SECONDARY OUTCOMES:
Change from baseline on tumor volume measured by enhanced pituitary Magnetic Resonance Imaging（MRI） | Up to 6 months
  Record the tumor volume from enhanced pituitary MRI on every 3 month follow-up visits
Change from baseline of visual field scale | Up to 6 months
  Record the Visual field scale on every 3 month follow-up visit, 0 = normal, no vision loss; 1 = one quadrant vision loss; 2 = two quadrants of vision loss; 3 = three quadrants of vision loss; 4 = four quadrants of vision loss but retain a central tubular vision; 5 = blind
Change from baseline of visual acuity | Up to 6 months
  Record the Visual acuity on every 3 month follow-up visit.

IPD SHARING:
Plan to Share IPD: No
The individual patient Data would not be shared to the third facility, but the sponsor hasn't decided whether to share the individual patient date to the other related studies hold by himself in the future.

REFERENCES:
- [Result] Mukherjee J, Majji D, Kaur J, Constantinescu CC, Narayanan TK, Shi B, Nour MT, Pan ML. PET radiotracer development for imaging high-affinity state of dopamine D2 and D3 receptors: Binding studies of fluorine-18 labeled aminotetralins in rodents. Synapse. 2017 Mar;71(3):10.1002/syn.21950. doi: 10.1002/syn.21950. Epub 2016 Nov 30. PMID 27864853
- [Result] Melmed S, Casanueva FF, Hoffman AR, Kleinberg DL, Montori VM, Schlechte JA, Wass JA; Endocrine Society. Diagnosis and treatment of hyperprolactinemia: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Feb;96(2):273-88. doi: 10.1210/jc.2010-1692. PMID 21296991
- [Result] Schonitzer V, Haasters F, Kasbauer S, Ulrich V, Mille E, Gildehaus FJ, Carlsen J, Pape M, Beck R, Delker A, Boning G, Mutschler W, Bocker W, Schieker M, Bartenstein P. In vivo mesenchymal stem cell tracking with PET using the dopamine type 2 receptor and 18F-fallypride. J Nucl Med. 2014 Aug;55(8):1342-7. doi: 10.2967/jnumed.113.134775. Epub 2014 Jul 14. PMID 25024426